CLINICAL TRIAL: NCT05141682
Title: A Phase I/II Clinical Trial Evaluating CC-486 in Patients With Relapsed/Refractory T-Cell Large Granular Lymphocytic Leukemia (T-LGLL)
Brief Title: Oral Azacitidine for the Treatment of Relapsed or Refractory T-cell Large Granular Lymphocytic Leukemia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jonathan Brammer (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor-Investigator, Jonathan Brammer, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-21018; NCI-2021-08491 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: T-Cell Large Granular Lymphocyte Leukemia
MeSH Terms: conditions — Leukemia, Large Granular Lymphocytic | interventions — Azacitidine; cc-486

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Oral Azacitidne) (Experimental): Patients will receive CC-486 orally (PO) D1-14 of a 28-day cycle, in a similar fashion to the QUAZAR study for a minimum of 4 cycles. Patients that achieve a response (CR or PR) will remain on study for a maximum of 12 months. Patients without a response at 4 months will come off the study.
  Interventions: Drug: Oral Azacitidine

INTERVENTIONS:
Drug: Oral Azacitidine — Given PO
  Other Names: CC-486

SUMMARY:
This phase I/II trial studies the best dose, possible benefits and/or side effects of oral azacitidine in treating patients with T-cell large granular lymphocytic leukemia that has come back (relapsed) or has not responded to previous treatment (refractory). Chemotherapy drugs, such as azacitidine, work in different ways to stop the growth of cancer cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety and maximum tolerated dose (MTD) of oral azacitidine (CC-486) in patients with symptomatic T-cell large granular lymphocytic leukemia (T-LGLL). (Phase I) II. To determine the overall response rate (complete response [CR] and partial response [PR]) of CC-486 in patients with T-LGLL. (Phase II)

SECONDARY OBJECTIVES:

I. Duration of response to CC-486. II. Progression-free survival. III. Rate of conversion from PR at 4 months to CR at 8 and 12 months. IV. Rate of molecular remission (T-cell receptor [TCR] clearance, STAT3 mutation clearance) at 4, 8, 12 months.

V. Effect of treatment on IL-15 promoter demethylation. VI. Effect of CC-486 on IL-15 promoter demethylation. VII. Safety of CC-486 in T-LGLL patients.

OUTLINE: This is a dose-escalation study.

Patients receive azacitidine orally (PO) on days 1-14. Treatment repeats every 28 days for 4 cycles in the absence of disease progression or unacceptable toxicity. Patients with PR or CR continue treatment for up to 8 additional cycles in the absence of disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Diagnosis of T-LGLL defined as: CD3+CD8+ cell population > 650/mm^3 and the presence of a clonal T-cell receptor (within 1 month of diagnosis). This also includes patients with rare T-LGLL variants include CD4+ T-LGLL, and gamma/delta T-LGLL which can be CD4- and CD8, though patients still must have an LGL cell population >500 cells/mm3 and the presence of a clonal T-cell receptor within 1 month of diagnosis or relapse. Note: patients with myelodysplastic syndrome (MDS)-like T-LGLL may be included with principal investigator (PI) approval even if CD3+CD8+ cell population is < 650/mm^3, though +TCR is required. Natural-killer (NK) large granular lymphocytic leukemia (LGL) is also permitted, provided there is a clonal NK-cell population noted with > 500 cells/mm^3
* Failed at least one line of frontline therapy; off treatment for at least 14 days or 5 half-lives, whichever is longer
* Require Treatment for T-LGLL (One or more required)

  * Symptomatic anemia with hemoglobin < 10 g/dL
  * Transfusion-dependent anemia
  * Neutropenia with absolute neutrophil count (ANC) < 500/mm^3
  * Neutropenia with ANC < 1500/mm^3 with recurrent infections
* Platelet count >= 50 x 10^9/L
* Serum creatinine =< 2 x the upper limit of normal (ULN)
* Total bilirubin =< 1.5 x ULN (patients with Gilbert's syndrome with a bilirubin > 1.5 x ULN permitted)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 1.5 x ULN
* Eastern cooperative oncology group (ECOG) performance status =< 2
* Men and women of reproductive potential must agree to follow accepted birth control methods for the duration of the study. Female subject is either post-menopausal or surgically sterilized or willing to use an acceptable method of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, condom with spermicide, or abstinence) for the duration of the study. Male subject agrees to use an acceptable method for contraception for the duration of the study
* Able to sign informed consent

Exclusion Criteria:

* Active Infection requiring ongoing anti-microbial treatment. Patients with human immunodeficiency virus (HIV), positive hepatitis B surface antigen or hepatitis C antibody will be excluded
* Concurrent immune-suppressive therapy (prednisone or equivalent up to 20 mg permitted to treat T-LGL symptoms, but must be weaned within one month of initiation of trial drug). Patients on stable, chronic prednisone =< 10 mg for rheumatologic/autoimmune conditions are exempted from this requirement. They may enroll on the study
* Active, concurrent malignancy unless deemed related to T-LGLL by PI
* Prior use of 5-azacytidine or decitabine
* Positive pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of oral azacitidine (CC-486) (Phase I) | Up to 4 cycles (1 cycle = 28 days)
Overall response rate (complete response [CR] + partial response [PR]) (Phase II) | Up to 3 years
  Assessed by the investigator based upon criteria derived from the ECOG 5998 and BNZ-1 clinical trials.

SECONDARY OUTCOMES:
Duration of response to CC-486 | Up to 3 years
Progression-free survival (PFS | Up to 3 years
Rate of conversion from PR at 4 months to CR at 8 months | From 4 months to 8 months
Rate of conversion from PR at 4 months to CR at 12 months | From 4 months to 12 months
Rate of molecular remission (T-cell receptor [TCR] clearance, STAT3 mutation clearance) | At 4 months
Rate of molecular remission (TCR clearance, STAT3 mutation clearance) | At 8 months
Rate of molecular remission (TCR clearance, STAT3 mutation clearance) | At 12 months
Rate of treatment-emergent adverse events | Up to 12 months
Degree of IL-15 promoter demethylation in responders versus non-responders | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Brammer, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center
Locations (2):
- United States (2):
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Virginia, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu